CLINICAL TRIAL: NCT02161120
Title: Effects of Traditional and Low-FODMAP Rye Bread in Irritable Bowel Syndrome.
Brief Title: Effect of Two Different Rye Bread Types in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oy Karl Fazer Ab (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BSTN-2014-rye
Record Dates: First submitted 2014-06-10; First posted 2014-06-11 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS, irritable bowel syndrome, functional gastrointestinal disorder, diet, bread, rye, FODMAP, microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens; Gastrointestinal Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional rye bread (Active Comparator): As part of habitual diet participants are expected to consume 100-200 grams of traditional Finnish rye bread daily
  Interventions: Other: Traditional Finnish rye bread
- Low-FODMAP rye bread (Experimental): As part of habitual diet participants are expected to consume 100-200 grams of low-FODMAP rye bread daily
  Interventions: Other: Low FODMAP rye bread

INTERVENTIONS:
Other: Traditional Finnish rye bread
  Arms: Traditional rye bread
Other: Low FODMAP rye bread
  Arms: Low-FODMAP rye bread

SUMMARY:
The purpose of this study is to evaluate if low-FODMAP (Fermented Oligo-, Di-, Monosaccharides And Polyols) rye bread is better tolerated in irritable bowel syndrome than commonly available traditional rye bread higher in FODMAP carbohydrates. The study also aims to investigate patients' compliance to rye bread regimen, potential changes is gut microbiota and hydrogen production during the test periods (a marker of large bowel fermentation of poorly absorbed carbohydrates).

ELIGIBILITY:
Inclusion Criteria:

* IBS according to Rome III criteria. Accepted sub-types include IBS-M, IBS-D and IBS-U
* Age 18-65 years
* Willing to use rye bread daily during the study periods

Exclusion Criteria:

* IBS-C (constipation dominant)
* Celiac disease
* IBD
* Major gastrointestinal operations like bowel gastric resection
* Non-treated hypo- or hyperthyroidism
* Alcoholism, severe depression, dementia, cancer or other diseases likely to severly impair the participants ability to conclude the protocol
* Regular (almost daily) use of NSAIDs, antibiotics or lactulose
* Linaclotide and other prescription medicines targeted specifically to IBS
* Pregnancy and lactation
* Follows currently strict low-FODMAP diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2014-04; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change is IBS symptoms by using IBS-SSS questionaire | 4 weeks

SECONDARY OUTCOMES:
IBS quality of life by using IBS QoL questionnaire | 4 weeks
Changes in specific IBS symptoms measured by 100 mm VAS scale | 4 weeks
Changes is intestinal microbiota evaluated by fecal samples | 4 weeks
Changes in hydrogen excretion evaluated by 6 hours breath test after standard rye bread breakfast | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Aava Medical Centre, Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Laatikainen R, Jalanka J, Loponen J, Hongisto SM, Hillila M, Koskenpato J, Korpela R, Salonen A. Randomised clinical trial: effect of low-FODMAP rye bread versus regular rye bread on the intestinal microbiota of irritable bowel syndrome patients: association with individual symptom variation. BMC Nutr. 2019 Mar 6;5:12. doi: 10.1186/s40795-019-0278-7. eCollection 2019. PMID 32153925